CLINICAL TRIAL: NCT03884114
Title: Assessment of Clinical Competence of Medical Students: a Comparison of High-fidelity Simulation, Serious Game and Multiple-choice Questions
Brief Title: Comparison of Three Modalities to Assess Clinical Competence of Medical Students
Acronym: SIMEVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilumens (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Ilumens0003
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Educational Problems
Keywords: technology-enhanced simulation; serious games; multiple choice questionnaires; medical education

STUDY DESIGN:
Intervention Model Description: All medical students are evaluated using a high-fidelity simulation environment, then using a serious game, then using multiple choice questionnaire, all on the same topic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All participants are evaluated on a scenario of pediatric asthma exacerbation using three different evaluation tools: (i) the simulation game EfficAsthme developed to train individuals on the management of pediatric asthma exacerbations; (ii) a MCQ on the same subject developed for the purpose of the study and (iii) HF-simulation, considered as the gold-standard for its enhanced realism.
  Interventions: Other: High-fidelity simulation; Other: Simulation game; Other: Multiple choice questionnaire

INTERVENTIONS:
Other: High-fidelity simulation — The first evaluation modality studied is high fidelity (HF) simulation. In our study, this modality is considered to be the gold-standard assessment method of clinical assessment, because HF simulation corresponds to the modality which reflects the best clinical competence in hospital settings. The HF pediatric manikin used (SimBaby), is able to reproduce all the signs of an asthma exacerbation (coughing, wheezing, tachypnea, chest indrawing, seesaw respiration, cyanosis). In the simulation room, participants can use the same items that those present in the simulation game (a glass of water, paracetamol, short acting beta-agonist, controller treatment (Fluticasone), an asthma spacer with a facial mask, saline nose drops to perform nasal irrigation, oral steroids in tablets (prednisone), and a phone).
Other: Simulation game — EfficAsthme is a simulation game used on a tablet computer. This simulation game was developed to train parents on the management of asthma exacerbations of their children. For the purpose of the study, EfficAsthme is diverted from its original use to assess students' clinical skills. The training scenario "A polluted atmosphere" is used in this study. Participants need to observe the signs presented by the child, and to determine the severity of the asthma exacerbation. From a menu on the right of the screen, the participant can choose several actions, especially to provide the short acting beta-agonist.
Other: Multiple choice questionnaire — The third evaluation modality corresponds to a multiple choice questionnaire (MCQ) including 15 questions. As for HF-simulation and the simulation game, the MCQ starts with the same briefing and continues with 15 questions regarding the management of a moderate asthma exacerbation.

SUMMARY:
This study, focusing on the management of pediatric asthma exacerbations, assesses the clinical skills of medical students using three different evaluation tools: (i) the simulation game "Effic'Asthme" developed to train individuals on the management of pediatric asthma exacerbations; (ii) a multiple choice questionnaire (MCQ) on the same subject developed for the purpose of the study and (iii) high fidelity (HF)-simulation, considered as the gold-standard for its enhanced realism.

Its objective is to determine which of the simulation game or the MCQ reflects the best the clinical competence of medical students evaluated on a HF simulator.

DETAILED DESCRIPTION:
The assessment of medical students' clinical competence has long been of concern to educational institutions. Objective structural clinical examination (OSCE) and assessments in high-fidelity (HF) simulation settings represent interesting evaluation modalities but are associated with huge costs, especially when they are used for large-scale standardized assessments. Multiple choice questionnaires (MCQ) remain the most common evaluation tool in medical schools.

Simulation games may represent an interesting compromise between the cheap but limited assessment allowed by MCQs, and the comprehensive but highly expensive assessment allowed by OSCE and HF simulation.

This study, focusing on the management of pediatric asthma exacerbations, assesses the clinical skills of medical students using three different evaluation tools: (i) the simulation game "Effic'Asthme" developed to train individuals on the management of pediatric asthma exacerbations; (ii) a MCQ on the same subject developed for the purpose of the study and (iii) HF-simulation, considered as the gold-standard for its enhanced realism.

Its objective is to determine which of the simulation game or the MCQ reflects the best the clinical competence of medical students evaluated on a HF simulator.

ELIGIBILITY:
Inclusion Criteria:

* medical students from Paris 5 University who meet the following criteria

  * Being in their fifth year of medical school
  * Having passed their pediatric exam in the previous 15 days
  * Willing to participate in the study

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
Items of the "asthma exacerbation performance score" | Baseline
  This score uses a scale designed for the purpose of the study, the "Asthma exacerbation performance score", ranging from 0 to 19, 19 being the highest rate meaning that all the actions were correctly performed (1 point per action correctly performed).
  This score will allow to calculate the degree of correlation calculated by Kappa coefficient for each action performed or answer provided, between the simulation game and the high fidelity simulation session on the one hand; and between the multiple choice questionnaire and the high fidelity simulation session on the other hand;
  Then, we will compare the median Kappa coefficients for each condition, and determine which of the multiple choice questionnaire or the simulation game reflects the best the clinical competence of medical students observed during a high-fidelity simulation session.

SECONDARY OUTCOMES:
The total score on the "asthma exacerbation performance score" | Baseline
  The total scores of this checklist will allow to calculate:
  * the degree of correlation of the scores using this checklist between the simulation game and the high-fidelity simulation session using spearman correlation,
  * the degree of correlation of the scores using this checklist between the simulation game and the multiple choice questionnaire using spearman correlation
  It will also allow to compare the median scores of the students between the three modalities of assessment (high fidelity simulation, simulation game and multiple choice questionnaire), and the dispersion of the scores between the three modalities.
The satisfaction of students using Likert-scales with each evaluation modality | Baseline
  The satisfaction of students with the simulation game, and with the multiple choice questionnaire, will be assessed using a questionnaire with Likert-scales.

CONTACTS AND LOCATIONS:
Overall Officials: David Drummond, MD, PhD, Principal Investigator — Université Paris Descartes
Locations (1):
- Université Paris Descartes, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
* Participants' characteristics anonymized
  * Participants' correct and incorrect actions and answers when evaluated on the 3 different modalities: multiple choice questionnaire, high-fidelity simulation and simulation game
Supporting Information: Study Protocol, SAP
Time Frame: From baseline to 2 years after completion of the study.
Access Criteria: Individual patient date, study protocol and statistical analysis plan will be available upon request to david.drummond@ilumens.org

REFERENCES:
- [Background] Norcini JJ, Swanson DB, Grosso LJ, Webster GD. Reliability, validity and efficiency of multiple choice question and patient management problem item formats in assessment of clinical competence. Med Educ. 1985 May;19(3):238-47. doi: 10.1111/j.1365-2923.1985.tb01314.x. PMID 4010571
- [Background] Drummond D, Delval P, Abdenouri S, Truchot J, Ceccaldi PF, Plaisance P, Hadchouel A, Tesniere A. Serious game versus online course for pretraining medical students before a simulation-based mastery learning course on cardiopulmonary resuscitation: A randomised controlled study. Eur J Anaesthesiol. 2017 Dec;34(12):836-844. doi: 10.1097/EJA.0000000000000675. PMID 28731928
- [Background] Adjedj J, Ducrocq G, Bouleti C, Reinhart L, Fabbro E, Elbez Y, Fischer Q, Tesniere A, Feldman L, Varenne O. Medical Student Evaluation With a Serious Game Compared to Multiple Choice Questions Assessment. JMIR Serious Games. 2017 May 16;5(2):e11. doi: 10.2196/games.7033. PMID 28512082
- [Derived] Fonteneau T, Billion E, Abdoul C, Le S, Hadchouel A, Drummond D. Simulation Game Versus Multiple Choice Questionnaire to Assess the Clinical Competence of Medical Students: Prospective Sequential Trial. J Med Internet Res. 2020 Dec 16;22(12):e23254. doi: 10.2196/23254. PMID 33325833
- See also: Site showing the simulation game "EfficAsthme" developed — http://sites-e-play.parisdescartes.fr/educasthma/efficasthme/